CLINICAL TRIAL: NCT01355003
Title: Quadrivalent Human Papillomavirus (Types 6, 11, 16, 18) Recombinant Vaccine (GARDASIL™) Post Marketing Surveillance Protocol
Brief Title: GARDASIL™ Post Marketing Surveillance in the Philippines (V501-077)
Status: Terminated | Type: Observational
Why Stopped: Merck Sharp & Dohme Corp (MSD) received exemption from PFDA on conduct of post-marketing surveillance (PMS) study
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: V501-077
Record Dates: First submitted 2011-05-16; First posted 2011-05-17 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Papillomavirus Infections
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Participants: Participants who were vaccinated with GARDASIL™ by their physician

SUMMARY:
This study will collect safety information on the use of GARDASIL™ in the Philippines.

ELIGIBILITY:
Inclusion Criteria:

* Received GARDASIL™

Ages: 9 Years to 46 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Data will be collected from physicians who prescribed GARDASIL™ and who voluntarily agree to provide information on their patients. Each physician can provide up to five reports corresponding to five patients.
Sampling Method: Non-Probability Sample
Enrollment: 1080 (Actual)
Dates: Start 2008-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events following any dose of vaccine | At least 30 days following any vaccine dose